CLINICAL TRIAL: NCT05068206
Title: A Multi-center, Randomized, Open-label Phase II Clinical Study to Evaluate the Efficacy and Safety of AK105 Plus Anlotinib and CapeOx, Anlotinib in Combination With CapeOx Versus Bevacizumab in Combination With CapeOx in the Fisrt-line Treatment of Unresectable Metastatic Colorectal Cancer
Brief Title: A Clinical Study to Compare the Efficacy and Safety of AK105 Plus Anlotinib and Capecitabine/Oxaliplatin (CapeOx) , Anlotinib Plus CapeOx, Bevacizumab Plus CapeOx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK105-II-04
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Unresectable Metastatic Colorectal Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK105+Anlotinib+CapeOx (Experimental): Treatment period (6 cycles):
  AK105 injection: intravenous drip on Day 1; Anlotinib hydrochloride capsule: oral administration, once daily(QD) ; Oxaliplatin for injection: intravenous infusion on Day 1; Capecitabine tablet:oral administration, twice daily (BID) .
  Maintenance period:
  AK105 injection: intravenous drip on Day 1; Anlotinib hydrochloride capsule: oral administration, once daily(QD) ; Capecitabine tablet:oral administration, twice daily (BID) . Every 3 weeks is as one cycle.Oxaliplatin is administered for 6 cycles, and AK105 can be administered continuously for 1 year but at most for 2 years. Other cases continue to be administered until the treatment termination event specified in the plan occurs.
  Interventions: Drug: AK105 injection; Drug: Anlotinib hydrochloride capsule; Drug: CapeOX
- Anlotinib+CapeOx (Experimental): Treatment period (6 cycles) Anlotinib hydrochloride capsule: QD orally; Oxaliplatin for injection: D1 intravenous infusion on Day 1; Capecitabine tablet: BID oral administration.
  Maintenance period:
  Anlotinib hydrochloride capsule: QD orally; Capecitabine tablet: BID oral administration. Every 3 weeks is as one cycle, and Oxaliplatin is administered for 6 cycles. Other cases continue to be administered until the treatment termination event specified in the plan occurs.
  Interventions: Drug: Anlotinib hydrochloride capsule; Drug: CapeOX
- Bevacizumab+CapeOx (Active Comparator): Treatment period (6 cycles):
  Bevacizumab D1 intravenous infusion; Oxaliplatin D1 intravenous infusion; Capecitabine BID oral administration.
  Maintenance period:
  Bevacizumab D1 intravenous infusion; Capecitabine BID oral administration. Every 3 weeks is as one cycle, and Oxaliplatin is administered for 6 cycles. Other cases continue to be administered until the treatment termination event specified in the plan occurs.
  Interventions: Drug: CapeOX; Drug: Bevacizumab

INTERVENTIONS:
Drug: AK105 injection — AK105 is programmed death 1（PD-1） monoclonal antibody
  Arms: AK105+Anlotinib+CapeOx
Drug: Anlotinib hydrochloride capsule — Anlotinib is small molecule multi-target tyrosine kinase inhibitor.
  Arms: AK105+Anlotinib+CapeOx; Anlotinib+CapeOx
Drug: CapeOX — CapeOX is Capecitabine+Oxaliplatin. Capecitabine is a kind of fluorouracil drug, and Oxaliplatin is a kind of platinum anticancer drug.
Drug: Bevacizumab — Bevacizumab is a recombinant human monoclonal antibody.
  Arms: Bevacizumab+CapeOx

SUMMARY:
A clinical study to compare the efficacy and safety of AK105 plus anlotinib and Capecitabine/Oxaliplatin (CapeOx) , anlotinib plus CapeOx, bevacizumab plus CapeOx. A total of 120 cases will be enrolled to the group.

ELIGIBILITY:
Inclusion Criteria:

* The subjects shall volunteer to join in the research and sign the informed consent under the good compliance.
* Aged: 18-75 (calculated on the date of signing informed consent); the physical status of Eastern cooperative oncology group 0~1; expected lifetime≥3 months.
* Unresectable and untreated metastatic colorectal adenocarcinoma patients diagnosed by histopathology Union for International Cancer Control (UICC) ,American Joint Committee on Cance( AJCC) tumor node metastasis staging system for colorectal cancer (8th edition in 2017) is clearly IV stage.
* Subjects who have not received systematic treatment for colorectal cancer before, including chemotherapy, targeted therapy and immunotherapy; Subjects with tumor recurrence or metastasis at least 6 months after the end of previous adjuvant or neoadjuvant chemotherapy.
* It can provide previously stored tumor tissue specimens or biopsy to collect tumor focus tissues for detecting programmed death 1 expression and kirsten rat sarcoma viral oncogene/neuroblastoma rat sarcoma viral oncogene mutation.
* According to RECIST 1.1 criterion, there is at least one measurable lesion. It is required that the selected target lesion has not received local treatment before, or the selected target lesion is located in the previous local treatment area, but it is determined as progressive disease by imaging examination.
* Good organ function (no blood transfusion, no hematopoietic stimulating factor, no infusion of albumin or blood products within 14 days before randomization).
* Female subjects of childbearing age should agree that contraceptive measures (such as abstinence, intrauterine device, contraceptive pills or condoms) must be used during the study and within 6 months after the end of the study; Serum pregnancy test was negative within 7 days before the study was enrolled, and it must be a non-lactating subject; Male subjects should agree that contraception must be used during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* 1) Combined diseases and medical history:

  1. Other malignant tumors have occurred or are currently suffering at the same time within 3 years. The following conditions can be included: cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invasive basement membrane)];
  2. Factors which affecting oral administration of drugs (such as inability to swallow, chronic diarrhoea and ileus, etc.);
  3. There is or tends to be gastrointestinal bleeding or perforation within 4 weeks before inclusion;
  4. Subjects with ulcerative colitis and Crohn's disease; Subjects with active inflammatory bowel disease within 4 weeks before inclusion;
  5. Uncontrollable pleural effusion and ascites requiring repeated drainage, and moderate and above hydropertcardium;
  6. Unmitigated toxic reactions above Common Terminology Criteria for Adverse Events S1 due to any previous treatment, excluding alopecia;
  7. Major surgical treatment, open biopsy or obvious traumatic injury were received within 28 days before inclusion (except tissue biopsy under gastrointestinal endoscope);
  8. Imaging(CT or MRI) showed that the tumor invaded large blood vessels or had unclear boundary with blood vessels;
  9. Subjects with hematemesis and hematochezia symptoms within 3 months before screening, and the daily bleeding volume is ≥ 2. 5 ml, or any bleeding event ≥ Common Terminology Criteria for Adverse Events S3, or subjects with any bleeding signs or medical history judged by researchers to be unsuitable for inclusion regardless of severity;
  10. There are unhealed wounds, ulcers or fractures;
  11. Arteriovenous thrombosis occurred within 6 months, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc;
  12. Subjects who have a history of psychotropic drug abuse and can't quit;
  13. Subjects with any severe and/or uncontrolled diseases, including:

Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after standard antihypertensive treatment); Suffering from unstable angina pectoris/ S2 or over cardiogenic chest pain; Myocardial infarction occurred within 12 months before randomization; S1or over heart failure (New York Heart Association (NYHA) grade); Restrictive cardiomyopathy; S2 or over atrioventricular block, arrhythmia that cannot be stably controlled by drugs [including QTc ≥ 450 ms (male) and QTc ≥ 470 ms (female)], and arrhythmia that may have potential influence on experimental treatment; Active infection (≥ Common Terminology Criteria for Adverse Events S2 infection); Decompensated cirrhosis, active hepatitis *; (* Active hepatitis (hepatitis B reference: HBsAg positive, and HBV DNA positive (> 2500 copies/ml or > 500IU/ml); Hepatitis C reference: HCV antibody positive, and HCV virus titer detection value exceeds the upper limit of normal value); Note: Subjects with positive hepatitis B surface antigen or core antibody and hepatitis C patients who meet the entry conditions need continuous antiviral treatment to prevent virus activation. ) Subjects with renal failure requiring hemodialysis or peritoneal dialysis; Have a history of immunodeficiency, including HIV positive or suffering from other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation; Diabetes mellitus is poorly controlled (fasting blood glucose (FBG) > 10mmol/L) Urine routine indicates that urine protein is ≥ + +, and it is confirmed that 24-hour urine protein quantity is > 1.0 g; Subjects who have a definite history of neurological or mental disorders, including epilepsy or dementia, and need treatment.

* 2) Tumor-related symptoms and treatment:

  1. Have received surgery (except previous diagnostic biopsy), radiotherapy, chemotherapy or other anti-cancer therapy within 4 weeks before inclusion (wahsout period is calculated from the end of the last treatment); Note: Those who have received local radiotherapy in the past can be enrolled if the following conditions are met: the end of radiotherapy is more than 4 weeks from the start of study treatment (brain radiotherapy is more than 2 weeks), and the target lesions selected in this study are not in the radiotherapy area; Or the target lesion is located in the radiotherapy area, but the progress has been confirmed;
  2. Within 2 weeks before joining the group, subjects who received ready-for-use traditional Chinese medicine (including Compound Mylabris Capsule, Kang'ai Injection, Kanglaite Capsule/Injection, Aidi Injection, Brucea javanica Oil Injection/Capsule, Xiaoaiping Tablet/Injection, Cinobufagin Capsule, etc.) with anti-tumor indications specified in National Medical Products Administration approved drug instructions;
  3. Subjects who have previously received anti-PD-1 or anti-PD-L1/PD-L2 preparations or other treatments acting on T cell co-stimulation targets or checkpoints;
  4. Previous postoperative adjuvant therapy containing anti-vascular or anti-epidermal growth factor receptor targeted drugs (including but not limited to bevacizumab, cetuximab, panitumumab, aflibercept, regorafenib, etc.)
  5. Central nervous system metastasis with symptoms or symptoms control time less than 2 months;
* 3) Research therapy related:

  1. Vaccination history of live attenuated vaccine within 28 days before enrollment or plan to vaccinate live attenuated vaccine during the study period;
  2. Subjects who are known to be allergic to research drugs or excipients, or allergic to similar drugs;
  3. Active autoimmune diseases requiring systemic treatment (such as the use of disease-relieving drugs, corticosteroids or immunosuppressants) occurred within 2 years before enrollment. Alternative therapies (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatment;
  4. Diagnosed as immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose > 10mg/day prednisone or other equivalent hormone), and continuing to be used within 2 weeks after the first administration;
* Participated in clinical trials of other anti-tumor drugs within 4 weeks before joining the group (washout period was calculated from the end of the last treatment);
* According to the researcher's judgment, there are accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study, or there are other reasons why the subjects are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival(PFS) | up to 8-10 months
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, the time between the beginning of randomization and the first occurrence of objective disease progression or recurrence or death from various causes (whichever occurs first).
Overall survival (OS) | up to 20-30 months
  Refers to the time between random grouping and death caused by various causes.
Objective remission rates(ORR) | up to 30 months
  Percentage of subjects with complete remission (CR) or partial remission (PR) as determined by RECIST 1.1.
Disease Control Rate (DCR) | up to 30 months
  Percentage of subjects with CR, PR, or disease stabilization (SD) at 6 weeks or more as determined by RECIST 1.1.

SECONDARY OUTCOMES:
Duration of disease remission (DOR) | up to 20-30 months
  For subjects whose best remission is CR or PR, it is defined as from the date when tumor remission is first recorded to the date when disease progression is first recorded or the date of death from any cause (whichever occurs first).

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yixian Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Scinece and Technology, Luoyang, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality